CLINICAL TRIAL: NCT07291635
Title: A Randomized, Observer-Blind, Adaptive, Active Comparator-Controlled, Dose-Ranging, Multicenter, Safety, Tolerability, and Immunogenicity Phase 1/2 Study of a Plant-Based Seasonal Recombinant Trivalent VLP Influenza Vaccine in Adults 18 Years of Age and Older
Brief Title: Phase 1/2 Study of a Plant-Based Seasonal Recombinant Trivalent VLP Influenza Vaccine
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aramis Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP-sFLUVLP-001
Record Dates: First submitted 2025-11-26; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1 (18-64): 15 μg (Experimental)
  Interventions: Biological: Recombinant Influenza vaccine candidate
- Group 2 (18-64): 30 μg (Experimental)
  Interventions: Biological: Recombinant Influenza vaccine candidate
- Group 3 (18-64): 60 μg (Experimental)
  Interventions: Biological: Recombinant Influenza vaccine candidate
- Group 4 (18-64): STD TIV (Active Comparator)
  Interventions: Biological: Commercial Influenza vaccine
- Group 5 (65+): 30 μg (Experimental)
  Interventions: Biological: Recombinant Influenza vaccine candidate
- Group 6 (65+): 60 μg (Experimental)
  Interventions: Biological: Recombinant Influenza vaccine candidate
- Group 7 (65+): HD TIV (Active Comparator)
  Interventions: Biological: Commercial Influenza vaccine

INTERVENTIONS:
Biological: Recombinant Influenza vaccine candidate — Plant-Based Seasonal Recombinant Trivalent TVLP Influenza Vaccine
  Arms: Group 1 (18-64): 15 μg; Group 2 (18-64): 30 μg; Group 3 (18-64): 60 μg; Group 5 (65+): 30 μg; Group 6 (65+): 60 μg
Biological: Commercial Influenza vaccine — Influenza vaccine commercially available on the Canadian market
  Arms: Group 4 (18-64): STD TIV; Group 7 (65+): HD TIV

SUMMARY:
This Phase 1/2 study is intended to assess the safety, tolerability, and immunogenicity of recombinant TVLP in adults 18-64 and 65 years of age and above and to confirm the dose(s) to be developed further in these two age cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have read, understood, and signed the informed consent form (ICF) prior to participating in the study; participants must also commit to complete study-related procedures and communicate with the study staff at visits and by phone during the study.
2. Participants must be 18 years of age and older at the Vaccination visit (Visit 2).
3. Participant must have a body mass index (BMI) ≤ 39 kg/m2 at the Vaccination visit (Visit 2).
4. Participants are considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study.
5. Participants cannot be living in an institutionalized setting (e.g. not living in rehabilitation centres or assisted living facilities; living in an elderly community like independent senior housing is acceptable), must be in good general health, and have no acute or evolving medical problems prior to study participation and no clinically relevant abnormalities that could jeopardize participant safety or interfere with study assessments, as assessed by the Principal Investigator or sub-Investigator (thereafter referred as Investigator) and determined by medical history, physical examination, serology, clinical chemistry and haematology tests, urinalysis, and vital signs. Investigator discretion will be permitted with this inclusion criterion.

Exclusion Criteria:

1. According to the Investigator's opinion, significant acute or chronic, uncontrolled medical or neuropsychiatric illness.
2. Any confirmed or suspected current immunosuppressive condition or immunodeficiency, including cancer, human immunodeficiency virus infection, hepatitis B or C (participants with a history of cured hepatitis B or C infection without any signs of immunodeficiency at present time are allowed). Investigator discretion is permitted with this exclusion criterion.
3. Participant is pregnant or lactating.
4. Participants who plan to become pregnant during the study period. Participants of child-bearing age who are currently or who become sexually active during the study should be willing to use effective birth control for the duration of the study. Participants of childbearing potential will undergo pregnancy testing at the screening visit and on Day 0 prior to vaccination.
5. Current autoimmune disease requiring systemic treatment (such as rheumatoid arthritis, systemic lupus erythematosus or multiple sclerosis). Investigator discretion is permitted with this exclusion criterion, and participants may be eligible to participate with appropriate written justification in the source document (i.e. participants with a history of autoimmune disease who are disease-free without treatment for three years or more, or on stable thyroid replacement therapy, mild psoriasis [i.e. a small number of minor plaques requiring no systemic treatment], etc.).
6. Administration of any non-influenza vaccine within 30 days prior to the Vaccination visit (Visit 2); planned administration of any vaccine up to Day 28 of the study. Immunization on an emergency basis during the study will be evaluated on case-by-case basis by the Investigator.
7. Administration of influenza vaccine within four months prior to the Vaccination visit (Visit 2).
8. Planned administration of influenza vaccine (other than the study vaccine) for six months post-administration or roll-out of the follow-year's seasonal influenza vaccination campaign: whichever comes first.
9. Use of any investigational or non-registered product within 30 days or five half-lives, whichever is longer, prior to the Vaccination visit (Visit 2) or planned use during the study period. Participants who are in a prolonged post-administration observation period of another investigational or marketed drug clinical study, for which there is no ongoing exposure to the investigational or marketed product and all scheduled on-site visits are completed, will be allowed to take part in this study, if all other eligibility criteria are met.
10. Administration of any medication or treatment that may alter the vaccine immune responses.
11. History of possible allergic reaction to any of the constituents of TVLP, any components of licensed vaccines, egg, or tobacco, based on the PI's assessment.
12. History of anaphylactic allergic reactions to plants or plants components (including fruits and nuts).
13. Participants with a history of Guillain-Barré Syndrome.
14. Use of prophylactic medications (e.g. antihistamines [H1 receptor antagonists], nonsteroidal anti-inflammatory drugs [NSAIDs], systemic and topical glucocorticoids, non-opioid and opioid analgesics) within 24 hours prior to the Vaccination visit (Visit 2) to prevent or pre-empt symptoms due to vaccination.
15. Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at the injection site that may interfere with injection site reaction rating. Investigator discretion will be permitted with this exclusion criterion.
16. Participants identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study, or any employees of Aramis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Immediate AEs | 30 minutes
  Percentage, intensity, and relationship to vaccination of immediate AEs (30 minutes post-vaccination)
Solicited local and systemic AEs | 7 days
  Percentage, intensity, and relationship to vaccination of solicited local and systemic AEs (for seven days following study vaccine administration)
Unsolicited AEs | 28 days
  Percentage, intensity, and relationship of unsolicited AEs, including TEAEs, for 28 days following study vaccine administration
Urine, haematological and blood biochemistry values | Screening and Day 3
  Number and percentage of participants with normal and abnormal, clinically significant urine, haematological and blood biochemistry values, and urinalysis at Screening visit and D3 (Phase 1 participants only)
Deaths, SAEs, AEs leading to withdrawal, TEAEs | 182 days
  Occurrences of deaths, SAEs, AEs leading to withdrawal, TEAEs, AESIs, NOCDs, and SUSARs up to the end of the study (D182)
HI antibody response (GMT) | Day 0 and Day 28
  HI antibody response (GMT) induced in TVLP Groups versus commercial comparator Groups against the homologous influenza strains on D0 and D28

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ward, MD, Study Chair — McGill University

IPD SHARING:
Plan to Share IPD: Undecided